CLINICAL TRIAL: NCT01645137
Title: Effectiveness Of Osteopathic Manipulative Treatment In Neonatal Intensive Care Units: A Multicenter Randomized Clinical Trial
Brief Title: Effectiveness Of Osteopathic Manipulative Treatment In NICU: A Multicenter Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Collaborators: Italian Academy of Traditional Osteopathy - AIOT (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Multi-NE-O
Record Dates: First submitted 2012-07-15; First posted 2012-07-20 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Prematurity
Keywords: prematurity; OMT; complementary and alternative medicine; neonates; length of stay
MeSH Terms: conditions — Premature Birth | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- OMT (Experimental): patients under usual medical care plus osteopathic treatment
  Interventions: Other: osteopathic manipulative treatment
- control (Other): patients under usual medical care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: osteopathic manipulative treatment — Patients from this group received osteopathic treatments twice a week for the entire length of stay in the unit.
  Arms: OMT
Other: Usual care — Patients from control group received standard care plus osteopathic evaluation only, according to the same schedule as the study group.
  Arms: control

SUMMARY:
The use of complementary and alternative medicine in neonatal ward has been steadily rising during the last decade. This integrated medicine approach has been shown to be helpful to improve neonatal health care. Osteopathic manipulative treatment (OMT) has been applied to premature infants to reduce the length of stay and to cope with clinical complications. Results from previous studies documented the positive association between OMT and shorter period of hospitalisation as well as improvement of clinical conditions. The aim of this nationwide multicenter study is to demonstrate the effect of OMT on length of stay (LOS) in premature infants across 3 neonatal intensive care units (NICU).

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born at age between 29 and 37 weeks
* osteopathic treatment performed < 14 days after birth
* preterms born in the same hospital

Exclusion Criteria:

* Gestational age < 29 weeks
* Gestational age > 37 weeks
* First OMT performed after 14 days from birth
* genetic disorders
* congenital disorders
* cardiovascular abnormalities
* proven or suspected necrotized enterocolitis with or without gastrointestinal perforation
* proven or suspected abdominal obstruction
* pre/post surgery patients
* pneumoperitoneum
* atelectasis
* Newborn from an HIV seropositive/drug addicted mother
* respiratory disorders
* transferred to/from other hospital
* admitted for preterminal comfort care (defined as neither intubation nor cardio-respiratory resuscitation)

Ages: 29 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 690 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of days of LOS | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

SECONDARY OUTCOMES:
pre-post difference in weight gain | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
number of episodes of vomit | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
days to full enteral feeding | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
NICU costs | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
number of episodes of regurgitation | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
number of episodes of stooling | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Monza Hospital, Monza, Lombardy
  - Macerata Hospital, Macerata, The Marches
  - Pescara hospital, Pescara

REFERENCES:
- [Derived] Cerritelli F, Pizzolorusso G, Renzetti C, Cozzolino V, D'Orazio M, Lupacchini M, Marinelli B, Accorsi A, Lucci C, Lancellotti J, Ballabio S, Castelli C, Molteni D, Besana R, Tubaldi L, Perri FP, Fusilli P, D'Incecco C, Barlafante G. A multicenter, randomized, controlled trial of osteopathic manipulative treatment on preterms. PLoS One. 2015 May 14;10(5):e0127370. doi: 10.1371/journal.pone.0127370. eCollection 2015. PMID 25974071
- [Derived] Cerritelli F, Pizzolorusso G, Renzetti C, D'Incecco C, Fusilli P, Perri PF, Tubaldi L, Barlafante G. Effectiveness of osteopathic manipulative treatment in neonatal intensive care units: protocol for a multicentre randomised clinical trial. BMJ Open. 2013 Feb 20;3(2):e002187. doi: 10.1136/bmjopen-2012-002187. Print 2013. PMID 23430598
- See also: Related Info — http://www.ebom.it
- See also: Related Info — http://www.aiot.edu